CLINICAL TRIAL: NCT04301479
Title: Low Dose Corticosteroid Infusion in Vasoplegia After Cardiac Surgery (CORTIVAS-CS): a Prospective Randomized Double-blinded Clinical Trial
Brief Title: Low Dose Corticosteroid Infusion in Vasoplegia After Cardiac Surgery (CORTIVAS-CS)
Acronym: CORTIVAS-CS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Principal Investigator, Filomena R B G Galas, Associate Professor of Anesthesiology at University São Paulo Medical School, Instituto do Coracao
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: InCor - HCFMUSP
Record Dates: First submitted 2020-02-27; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Vasoplegia; Cardiac Surgery
Keywords: vasoplegia; cardiac surgery; steroids
MeSH Terms: conditions — Vasoplegia | interventions — Hydrocortisone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroid (Active Comparator): Patients assigned for steroid group will receive 200 mg of hydrocortisone diluted in 120 mL of saline at an infusion rate of 5mL/hr for 3 days or shock reversal, defined by systolic arterial pressure > 90 mmHg for 12 hours after vasopressor weaning without fluid expansion.
  Interventions: Drug: hydrocortisone sodium succinate
- Control (Placebo Comparator): Patients assigned for control group will receive 120 mL of saline solution at a rate of 5mL/hr for 3 days or shock reversal, defined by systolic arterial pressure > 90 mmHg for 12 hours after vasopressor weaning without fluid expansion.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: hydrocortisone sodium succinate — Steroid group will receive 200 mg of hydrocortisone diluted in 120 mL of saline at an infusion rate of 5mL/hr for 3 days or shock reversal
  Arms: Steroid
Drug: Saline — Control group will receive 120 mL of saline solution at a rate of 5mL/hr for 3 days or shock reversal
  Arms: Control

SUMMARY:
Vasoplegia is an important determinant for adverse postoperative outcome and is observerd in 5% to 54% of patients undergoing cardiac surgery using cardiopulmonary bypass (CPB).

Postoperative vasoplegia is defined as a state with low systemic vascular resistance despite a normal or high cardiac output, and the need for vasopressor therapy.

Steroids attenuate the inflammatory response to cardiopulmonary bypass,but their effect on clinical outcomes is uncertain.

This is a double-blinded, randomized, clinical trial designed to determine the efficacy of low dose corticosteroid infusion in vasopressor free-days in vasoplegia after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with cardiopulmonary bypass
* Norephinerine treatment in ICU with dose great or equal than 0,1 mcg/kg/min to maintain or restore a MAP over 70 mmHg for at least 30 minutes within 24 hours after surgery

Exclusion Criteria:

* Preoperative vasopressor use (within 72 hours prior to surgery)
* Preoperative steroids use (within 7 days prior to surgery)
* Presence of ventricular assist device other than intraaortic ballon pump
* Transplant procedures
* Emergency procedures
* Aortic repairs
* Congenital procedures
* Endocarditis
* Bacterial or fungal infection in the preceding 30 days
* Active neoplasia
* Pregnancy
* Recent history of gastrointestinal bleeding
* Allergy or intolerance to steroids
* Participation in other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Vasopressors-free days | 30 days
  Days free of vasopressors up to day 30

SECONDARY OUTCOMES:
30 days mortallity | 30 days
  The number of deaths within 30 days of surgery
ICU length of stay | 30 days
  Duration in days from the date of the ICU admission to the date of ICU discharge
Infection complication | 30 days
  Rate of new infection or septic shock within 30 days after randomization
Acute myocardial infarction | 30 days
  We will compare the incidence of acute myocardial infarction between groups within 30 days after randomization
Atrial fibrillation | 30 days
  We will compare the incidence of atrial fibrillation between groups within 30 days after randomization

OTHER OUTCOMES:
Duration of mechanical ventilation | 30 days
  Duration in hours from the intraoperative intubation to postoperative extubation
Post-operative length of stay | 30 days
  Post-operative LOS is the duration in days from the date of the end of surgery to the date of discharge from hospital.
Mesenteric ischemia | 30 days
  We will compare the atrial fibrillation between groups within 30 days after randomization
Acute respiratory distress syndrome | 30 days
  We will compare the incidence of acute respiratory distress syndrome between groups within 30 days after randomization
Stroke | 30 days
  We will compare the incidence of stroke between groups within 30 days after randomization
Hyperglycemia | Up to 72 hours
  Peak of capillary blood glucose glycemia up to 72 hours after the start the protocol solution
180 days mortallity | 180 days
  The number of deaths within 180 days of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Incor - Heart Institute - University of Sao Paulo, São Paulo, Brazil